CLINICAL TRIAL: NCT06701019
Title: Exploring and Understanding Female Breast Health Referral Behavours in Primary Care: A Qualitative Interview/Focus Group Study
Brief Title: Exploring Breast Referral Behaviours in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); CoppaFeel (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sponsor ref 24068; IRAS project ID: 334924 (Other: Health Research Authority)
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Female
Keywords: breast; qualitative; primary care; patient; female

STUDY DESIGN:
Intervention Model Description: All participants will be asked via email for their medical history/status and demographic information.
  Participants will either be involved in an online semi-structured interview or focus group discussion (FGD). Note: they may allocated to a FGD where they share common characteristics with other participants (eg, they are younger women or presented at their GP practice with non-lump symptoms). However, if the participants prefer to be interviewed instead, the student will accommodate this option.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Data collection (Other): Semi-structured interview or focus group discussion.
  Interventions: Other: Semi-structured interview/focus group discussion

INTERVENTIONS:
Other: Semi-structured interview/focus group discussion — All participants will be asked via email for their medical history/status and demographic information.
  Participants will either be involved in online semi-structured interview or focus group discussion (FGD). Note: they may allocated to a FGD where they share common characteristics with other participants (eg, they are younger women or presented at their GP practice with non-lump symptoms). However, if the participants prefer to be interviewed instead, the student will accommodate this option.

SUMMARY:
The study will explore the experiences of women going to see their GP with breast-related health concerns and will involve finding out more about factors which may help and hinder them getting referred to a specialist for suspected breast cancer. As well as considering implications for further research, the study aims to inform clinical practice in terms of potential improvements to related medical education and the development of tools that could be introduced/refined for enhancing GP referrals in this area.

Breast cancer is the most diagnosed cancer amongst UK women, with incidence rates increasing by around a quarter since the early 1990s. It accounts for 30% of all female diagnosed cancers and causes around 11,500 deaths in the UK annually. Early detection is key as stage at diagnosis is the most important predictor of health outcome and most cancers are diagnosed after symptomatic patients see their GP. This highlights the pivotal role of primary care with managing breast-related abnormalities in a timely and appropriate manner. Little is currently known about the research area, particularly from a qualitative standpoint.

Adult females who have been referred to secondary care by their GP because of a breast health concern will be eligible to take part in the study. Participants will mainly be recruited through the Nottingham Breast Institute, East Midlands GP surgeries, and the study funder's digital/online influencer channels. Participants will be involved in semi-structured interviews or focus groups, with the data collection phase expected to take around six months. The study is funded by breast health awareness charity, Coppafeel!.

The findings of a systematic review and analysis of breast cancer-related online support group messages, focusing on the experiences relating to women seeing their GP with breast-health issues (also being undertaken by the researcher), will also be used to triangulate and inform study findings.

DETAILED DESCRIPTION:
Exploratory, cross-sectional, retrospective semi-structured interview and focus group study across multi-centres.

Objectives:

* To find out about the factors women perceive as those which hindered and/or facilitated participants' referral to a breast clinic for further investigation, and how and why the female patients believe these occurred.
* To look at improvements/changes the participants believe could be implemented to improve the related management of their health, particularly from a medical education perspective.

Settings:

Interviews/focus groups will be held online wherever possible using the following to reach potential participants:

* New referral clinics at the Nottingham Breast Institute at Nottingham City Hospital
* NIHR 'research initiative site' GP practices across the East Midlands which elect to get involved as participant identification centres; and
* The funder's (CoppaFeel!) digital communications channels and those of its ambassadors/social media influencers to reach potential participants.

Number of participants:

Up to 40 participants may be recruited but the concept of information power will be used to inform actual sample size. The participants will be women who have been to see their GP with breast-related health issues/symptoms.

Interventions:

* Requesting responses to related medical history/status and demographic questions in advance of the related substantive interview or focus group discussion (once per participant) - approx. 30 mins
* One online semi-structured interview or focus group discussion per participant - approx. 1 hour.

Duration of study:

* Overall: six months (to start soon as all necessary approvals are in place)
* Per participant: up to three months.

Method of analysis:

Data collected will be examined using inductive thematic analysis. This analytical approach allows themes, patterns and meanings to be generated from the data, and in the process, help identify factors which participants perceive as helping or hindering their breast referral to secondary care among patients and primary care healthcare professionals; and why, and how, these occurred.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender females (assigned to the female sex at birth)
* Aged 18 years and over (no upper age limit)
* Have/had breast-related health concerns regardless of breast cancer diagnosis
* Have presented their symptoms initially in a primary care setting rather than having been alerted to potential issues during routine breast screening
* Been referred from primary care within the previous year
* Be using the NHS healthcare system in either England or Wales.

Exclusion Criteria:

* Females who would need a language translator to take part in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Barriers and facilitators to referral measured via data collected from a semi-structured interview or focus group discussion with up to 40 participants | From enrolment to data collection up to 3 months
  The factors women perceive as those which hindered and/or facilitated participants' referral to a breast clinic for further investigation, and how and why the female patients believe these occurred.

SECONDARY OUTCOMES:
Suggested health management improvements measured via data collected from a semi-structured interview or focus group discussion with up to 40 participants | From enrolment to data collection up to 3 months
  Improvements/changes the participants believe could be implemented to improve the related management of their health, particularly from a medical education perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To comply with the Data Protection Act, personal data will be deleted as soon as possible after it is no longer needed for the study and at the latest by six months of the end of the study. However, if participants agree, their contact details will be kept so as to send them the findings of the study and to contact them about participating in future research studies.